CLINICAL TRIAL: NCT04150419
Title: Evaluation of the Effectiveness of a Therapeutic Program for the Attentional Re-training of Chronic Pain Patients: Feasibility of E-care
Brief Title: Attentional Re-training for Chronic Pain Patients
Acronym: ABCD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RC18_0361
Record Dates: First submitted 2019-10-17; First posted 2019-11-04 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pelvic Perinal Pain
Keywords: Attentional bias modification training; chronic pelvi-perinal pain.
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1 (Experimental)
  Interventions: Other: Group 1
- G2 (Experimental)
  Interventions: Other: Group 2
- G3 (Active Comparator)
  Interventions: Other: Group 3 (control group)

INTERVENTIONS:
Other: Group 1 — Attentional training to avoid threatening, negative or pain-related information.
  Arms: G1
Other: Group 2 — Attention training for vigilance for positive emotional information.
  Arms: G2
Other: Group 3 (control group) — Neutral attentional training (control group).
  Arms: G3

SUMMARY:
Hyper-vigilance, focusing, avoidance are part of the vocabulary used by the clinician who deals with chronic pain. These notions refer to the functioning and dysfunction of so-called "selective" attention. These "selective attentional biases" are believed to be responsible, in part, for the development and maintenance of negative pain-related thoughts (such as catastrophic thoughts), inappropriate behaviours (such as inactivity and fear of movement) and unpleasant emotions (such as stress or anger). In addition, they would also be a powerful indicator of the onset of post-operative pain and could limit the effectiveness of therapeutic management. Therapeutically, attention bias can be "managed" through attentional re-training techniques (ABMs) that teach patients to direct their attention differently. These techniques have been widely validated in anxious or addictive populations but have never been used to date in chronic pain patients. This home-based attention bias management (e-retraining) would represent, for chronic pain patients, an additional tool aimed not only at reducing their pain but also at achieving other associated factors such as anxiety, stress, catastrophic thoughts, avoidance behaviours and quality of life.

DETAILED DESCRIPTION:
After obtaining the patients' agreement, they will be randomized in one of the 3 experimental groups:

* G1: Attentional training to avoid threatening, negative or pain-related information.
* G2: Attention training for vigilance for positive emotional information.
* G3: neutral attentional training (control group).

The study will be conducted from the patient's home via a connection to the protected site of the Nantes University Hospital. The various questionnaires will be completed from the secure site of the Nantes University Hospital and the computerized experimental tasks will be carried out using the Inquisit software (WEB version at home).

The study will begin with an evaluation of the patients' attention and psychological processes (completion of questionnaires + 2 attention tasks), during a follow-up visit to the urology department of the University Hospital of Nantes.

Then, an 8-week attentional re-training program (2 training sessions per week) will be proposed.

At the end of the 8 weeks, an evaluation (Questionnaires + attention tasks) will be offered to patients always from home.

Finally, a final evaluation, 4 weeks after the end of the re-training, will always be proposed from the patient's home.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain patients, i.e., chronic pain that has been ongoing for more than 3 months.
* Patient follow-up in the urology department of the University Hospital of Nantes
* Age between 18 and 65
* Good understanding of French, able to read and write.
* Serve correctly and painlessly with both hands
* Affiliated with a social security system
* Signed consent
* With internet access.

Exclusion Criteria:

* Current and unstable psychiatric (mood disorders, anxiety disorders) and addictive (substance use disorders, alcoholic or otherwise, excluding nicotine) disorders.
* Does not use both hands properly and painlessly
* Depression (BDI-II ≤18)
* Patient under guardianship, curatorship or judicial protection
* Pregnant or breastfeeding woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of a therapeutic program for attentional re-training on the painful feelings of patients with chronic pelvic-perineal pain. | 3 months
  Variation in pain assessed from the numerical scale. The Numerical Pain Rating Scale measures the perception of pain intensity with an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Quistrebert-Davanne, PhD, Principal Investigator — Nantes University Hospital Nantes
Locations (1):
- CHU Nantes, Nantes, France